CLINICAL TRIAL: NCT04076358
Title: A Tablet-based Simple Walking Intervention to Improve Self-management of Arthritis Fatigue
Brief Title: A Tablet-based Simple Walking Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Jeungok Choi, Associate professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-4832
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Arthritis; Fatigue
Keywords: arthritis, fatigue
MeSH Terms: conditions — Arthritis; Fatigue

STUDY DESIGN:
Intervention Model Description: The study uses an experimental pre- and post-test repeated measures design. Those satisfying the inclusion and exclusion criteria are randomly assigned to the intervention (Tab-CBI, n=12) or comparison group (n=12).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tab-CBI (Experimental): The Tab-CBI group receives a tablet preloaded with the Tab-CBI application and an accelerometer. During the study period, the participants have four weekly educational sessions plus one booster session by the research assistant through a videoconferencing tool. The educational modules were developed based on the principles of cognitive behavioral therapy. The key elements of the modules include activity-pacing, adjustment of goal-setting to the current physical condition, setting priorities and structured planning of a simple walking activity and time off, and cognitive restructuring of activity demands (see attached, outline of education modules).
  Interventions: Behavioral: Tab-CBI
- Usual Care (No Intervention): The usual care group receives Arthritis related fatigue management which are currently offered to the participants at the recruitment sites. Participant are also instructed to maintain usual activity during the study period. The control group participants also receive an accelerometer to count steps, but without a tablet.

INTERVENTIONS:
Behavioral: Tab-CBI — Participants receive a tablet preloaded with Tab-CBI application and an accelerometer.
  Arms: Tab-CBI

SUMMARY:
The purpose of this project is to pilot test the effect of a tablet-based cognitive behavioral intervention (Tab-CBI) application on older adults' a) daily steps, b) fatigue level, c) self-efficacy, and d) quality of life at Week 1 (baseline), Week 4 (intervention completion), Week 6 (booster), Week 8 (follow-up #1), and Week 10 (follow-up #2) in a sample of 24 older adults.

The investigators hypothesize that (a) individuals receiving Tab-CBI will have increased daily step counts, decreased fatigue level, greater perception of self-efficacy and quality of life than those receiving current RA fatigue management, and that (b) the effects will be sustained up through 4 weeks of follow-ups after the intervention completion.

DETAILED DESCRIPTION:
The study uses an experimental pre- and post-test repeated measures design. After eligible participants sign an informed consent form, the participants will be screened for inclusion and exclusion criteria using two surveys (PROMIS Fatigue-8a, Mini-Cog) and verbally asking about age, presence of Arthritis diagnosis, Wi-Fi availability, engagement of regular exercise, presence of any non-ambulatory condition that limits walking.

Those satisfying the inclusion and exclusion criteria are randomly assigned to the intervention (Tab-CBI, n=12) or comparison group (n=12). The Tab-CBI group receives a one-on-one introductory session which covers details about the study purpose and procedures, description of Tab-CBI, and instructions of how to operate a tablet, an accelerometer, and a videoconferencing tool. At the end of the session, participants are given a tablet preloaded with the Tab-CBI application and an accelerometer. During the study period, the participants will receive four weekly educational sessions plus one booster session at 2 weeks after the intervention conclusion. The educational modules were developed based on the principles of cognitive behavioral therapy. The key elements of the modules include activity-pacing, adjustment of goal-setting to the current physical condition, setting priorities and structured planning of a simple walking activity and time off, and cognitive restructuring of activity demands. Participants will record daily which steps taken by syncing the accelerometer to the tablet.

The comparison group receives fatigue management which are currently offered to the patients and will be instructed to maintain usual activity during the study period. The control group participants also receive an accelerometer to count steps, but without a tablet.

Participants in both groups take surveys for four outcomes (dally steps, fatigue, perceived self-efficacy, and perceived quality of life) and four potential covariate measures (pain, depression, sleep, and comorbidity) through a tablet computer (for intervention group) or paper-based surveys (for comparison group). Data are collected at Week 1 (baseline), Week 4 (intervention completion), Week 6 (booster), Week 8 (follow-up #1), and Week 10 (follow-up #2).

ELIGIBILITY:
Inclusion Criteria:

* age >=50
* has greater than minimal fatigue scoring ≥17 on the PROMIS Fatigue Short Form v1.0 Fatigue-8a.
* self-reported diagnosis of Arthritis
* having Wi-Fi at home.

Exclusion Criteria:

* those who are currently engaging in regular exercise
* non-ambulatory or having a condition that would limit the ability to walk (e.g., foot deformity, lower extremity joint surgery in past 6 months, stroke, severe chronic obstructive pulmonary disease, etc.)
* overt delirium, dementia, or any conditions indicating deteriorating cognitive status as determined by the Mini-Cog

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
daily steps | 24 hours
  daily step counts measured by an accelerometer
Fatigue severity | past 1 week
  self-reported fatigue severity measured by PROMIS Fatigue-8a
perception of self-efficacy | 24 hours
  self-reported self-efficacy measured by PROMIS Short Form v1.0 Self-Efficacy for Managing Symptoms-8a
perceived quality of life | past 2 weeks
  self-reported perception of quality of life measured by WHOQOL

CONTACTS AND LOCATIONS:
Overall Officials: Jeungok Choi, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No